CLINICAL TRIAL: NCT00161824
Title: Single-blind, Randomized, Multicenter Comparison of FSME IMMUN NEW and ENCEPUR: Safety and Tolerability of Two Vaccinations in Healthy Volunteers Aged 16 to 65 Years.
Brief Title: Safety Study in Volunteers From 16 to 65 Years of Age: FSME IMMUN NEW vs. ENCEPUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 208
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-borne
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated)

SUMMARY:
The purpose of this study is to assess the safety of a vaccination schedule consisting of two vaccinations (21-35 days apart) with the tick-borne encephalitis (TBE) vaccine FSME-IMMUN NEW (5 consecutive lots) in comparison to another licensed TBE vaccine (Encepur® adults, with polygeline) (2 lots) in healthy volunteers aged 16 to 65 years.

ELIGIBILITY:
Inclusion Criteria:

Male and female volunteers were eligible for participation in this study if they:

* Were 16 years (from the 16th birthday) to 65 years (to the last day before the 65th birthday) old
* Were clinically healthy
* Had a negative pregnancy test at the first medical examination, if female and capable of bearing children
* Agreed to employ adequate birth control measures for the duration of the study, if female and capable of bearing children
* Provided written informed consent
* For volunteers under 18 years of age - written informed consent of the parents / guardian was available
* Agreed to keep a volunteer diary

Exclusion Criteria:

* History of any previous TBE vaccination
* History of TBE infection or show evidence of latent TBE infection (as demonstrated by screening ELISA > 126 VIEU/ml)
* History of allergic reactions, in particular to one of the components of the vaccine
* Previously received volume substitution with a product containing polygeline (stabilizer in ENCEPUR)
* Received antipyretics within 4 hours prior to the first TBE vaccination
* Suffer from a disease that cannot be effectively treated or stabilized
* Suffering from a disease (e.g. autoimmune disease) or were undergoing any form of treatment that could be expected to influence immunological functions
* Suffering from chronic, degenerative and/or inflammatory disease of the central nervous system
* Using any immunosuppressive drugs (e.g. local or systemic corticosteroids, chemotherapeutics)
* Had a known or suspected problem with drug or alcohol abuse (> 4 liters wine / week or equivalent level of other alcoholic beverages)
* Had donated blood or plasma within one month of the study start
* Had received banked blood or immunoglobulins within one month of study entry
* Known to be HIV positive (a special HIV test was not required for the purpose of the study)
* Suffering from a febrile illness at study entry
* History of vaccination against yellow fever and / or Japanese B encephalitis
* Participating simultaneously in another clinical trial
* If female: pregnant or breast feeding

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3800
Dates: Start 2001-10; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Romaszko, MD, Principal Investigator — PANTAMED sp. z o o.; Jerzy Brzostek, MD, Principal Investigator — Zespol Opieki Zdrowotnej w Debicy; Jerzy Dziduch, MD, Principal Investigator — Samodzielny Publiczny Zaklad Opieki Zdrowotnej Oddzial Pediatryczny; Krystnyna Jurowska, MD, Principal Investigator — Przedsiebiorstwo Uslug Medycznych "Centrum Medyczne Nowa Huta"; Marian Patrzalek, MD, Principal Investigator — Wojewodzki Szpital Dzieciecy Oddzial Obserwacyjno - Zakazny A; Krzysztof Sladek, MD, Principal Investigator — "Atopia" Diagnostyka i Leczenie Chorob Alergicznych i Ukladu Oddechowego; Ryszard Konior, MD, Principal Investigator — Szpital Jana Pawla II Oddzial Neuoinfekcji
Locations (7):
- Poland (7):
  - Zespol Opieki Zdrowotnej w Debicy, Dębica
  - Wojewodzki Szpital Dzieciecy Oddzial Obserwacyjno - Zakazny A, Kielce
  - "Atopia" Diagnostyka i Leczenie Chorob Alergicznych i Ukladu Oddechowego, Krakow
  - Przedsiebiorstwo Uslug Medycznych "Centrum Medyczne Nowa Huta", Krakow
  - Szpital Jana Pawla II Oddzial Neuroinfekcji, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Oddzial Pediatryczny, Lubartów
  - PANTAMED sp. z o.o., Olsztyn